CLINICAL TRIAL: NCT02945462
Title: The Safety and Efficacy of Using Bone Marrow-derived Mesenchymal Stem Cells in the Treatment of Erectile Dysfunction in Diabetic Patients
Brief Title: Bone Marrow Mesenchymal Stem Cells in Erectile Dysfunction (ED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Saddam Dmour, Researcher, University of Jordan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDUJCTC
Record Dates: First submitted 2016-10-17; First posted 2016-10-26 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- autologous mesenchymal stem cells (Experimental): Intervention:
  Autologous bone marrow derived stem cells will be injected twice intracavernously to enrolled erectile dysfunction patients
  Interventions: Biological: autologous mesenchymal stem cells

INTERVENTIONS:
Biological: autologous mesenchymal stem cells — Patients will be injected with autologous mesenchymal stem cells, intracavernously

SUMMARY:
Recovery of erectile function using bone marrow mesenchymal stem cells (MSCs) after in vitro expansion under restricted culturing conditions.

DETAILED DESCRIPTION:
Four diabetic male patients ranging from 25-65 years diagnosed with erectile dysfunction will be selected. This diagnosis is based on medical history, validated questionnaires, physical examinations, laboratory tests and specific diagnostic tests. Patients with any evidence of untreated hypogonadism, current urinary tract or bladder infection, clinically evident penile anatomical deformities, previous penile implant or penile vascular surgery, uncontrolled hypertension or hypotension, reported unstable Cardiovascular diseases, uncontrolled diabetes (HbA1c > 10%), or primary hyperlipidemia will be excluded. The investigators hypothesize that the intracavernous injection of stem cells will facilitate the recovery of erectile function resulting in satisfying clinical outcomes in patients.

This study was performed:

1. To test the safety of autologous intracavernous bone marrow mesenchymal stem cells.
2. To evaluate benefit for the patient concerning recovery of natural erection by performing detailed and specific diagnostic tests prior and post MSCs injection by a team from Jordan University Hospital and Cell Therapy Center in Jordan University.
3. To study the feasibility, indication criteria and application modalities of Bone marrow mesenchymal stem cells for further wider study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male patients ranging from 25 to 65 years.
2. Type 1 or type 2 diabetic patients with a personal history of diabetes ≥ 5 years.
3. History of chronic erectile dysfunction for at least six months.
4. HbA1c ≤ 10%.
5. Baseline International Index of Erectile Function (IIEF) score of < 26.
6. Not interested or able to use Phosphodiesterase type 5 inhibitor (PDE-5i) drug therapy and willing to forgo these treatments for the first 6 month period following study treatment.
7. Body mass index between 20 -30.
8. Willing to provide written informed consent, complete questionnaire, and to be available for all baseline treatment and follow up examinations required by protocol.

Exclusion Criteria:

1. Untreated hypogonadism or low serum total testosterone < 200 ng/dl.
2. Current urinary tract or bladder infection.
3. Any medical evidence of any infectious disease.
4. Clinically evident penile anatomical deformities (e.g., Peyronie's disease) or history of priapism.
5. Skin irritation, infection, wound, sore or disruption in the immediate areas of skin entry for penile injection.
6. Current or previous malignancy.
7. Patients with primary hyperlipidemia.
8. Use of any non study treatment for erectile dysfunction within 4 weeks of study treatment.
9. Lack of willingness to continue through 6 months after study treatment.
10. Any previous penile implant or penile vascular surgery.
11. Uncontrolled hypertension or hypotension (systolic blood pressure > 170 or < 90 mm Hg, and diastolic blood pressure > 100 or < 50 mm Hg).
12. Reported unstable cardiovascular disease (e.g., unstable angina, myocardial infarction within past 6 months, cardiac failure or life-threatening arrhythmia, congestive heart failure) or symptomatic postural hypotension within 6 months before screening.
13. Bleeding or clotting disorder, use of anticoagulant therapy.
14. Lab values for complete blood count, prothrombin time/ partial thromboplastin time/international randomized ratio (PT/PTT/INR), Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and creatinine falling outside the normal lab values.
15. Systemic autoimmune disorder.
16. Significant active systemic or localized infection.
17. Receiving immunosuppressant medications.
18. HbA1c > 10%.

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-09; Primary Completion 2015-11 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | six months
  Observation of any relevant adverse side effect resulting from the injection. Assessing the safety of autologous Mesenchymal Stem Cells injection

SECONDARY OUTCOMES:
Assessment the efficacy of intracavernous injection measured by SHIM/IIEF/EHS questionnaire | 18 months
  Assessing the therapeutic benefits of the injected Autologous Mesenchymal Stem Cells by Sexual Health Inventory for Men/ International Index for Erectile Function/ Erection Hardness Score (SHIM/IIEF/EHS) questionnaire.
  For every patient tests would be performed at baseline and repeated at 1,3, 6,12, and 18 months post-injection.
Evaluation the efficacy of intracavernous injection measured by Dynamic Infusion cavernosometry test. | 6 months
  Assessing the therapeutic benefits of the injected Autologous Mesenchymal Stem Cells by Dynamic Infusion Cavernosometry test at baseline and repeated at 6 months post injection.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Al Demour S, Adwan S, Jafar H, Alhawari H, Awidi A. Stem cell therapy in diabetic men with erectile dysfunction: a 24-month follow-up of safety and efficacy of two intracavernous autologous bone marrow derived mesenchymal stem cells injections, an open label phase 2 clinical trial. Basic Clin Androl. 2024 Jul 5;34(1):13. doi: 10.1186/s12610-024-00229-y. PMID 38965462